CLINICAL TRIAL: NCT06283628
Title: Comparative Effectiveness of Two Different Approaches to Radiofrequency Ablation of Lumbar Medial Branch Nerves
Acronym: LMB-RFA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Bunty Shah, Associate Professor, Department of Anesthesiology and Perioperative Medicine, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00023737
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-10

CONDITIONS: Lumbar Spondylosis
MeSH Terms: conditions — Spondylosis

STUDY DESIGN:
Intervention Model Description: The subjects with bilateral low back pain will undergo radiofrequency ablation of the lumbar medial branch nerves using one approach (traditional) on one side and different approach (parasagittal) on the other side. One arm will use the traditional approach on the left and the parasagittal approach on the right. The other arm will use parasagittal approach on the left and the traditional approach on the right,
Who Masked: Participant, Outcomes Assessor
Masking Description: We will do computer randomization for the sides for each approach for all the subjects. The subjects will be assigned numbers, and the particular procedural approach for each side will be concealed in the numbered envelopes. The numbers on the envelopes will correspond to the numbers assigned to the patients. The envelopes will be opened by a treating physician in the procedure room. The patient and the assessor (who will not be the treating physician) will not know which procedural approach was used for the sides.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subjects with traditional approach on the right side and parasagittal approach on the left side. (Active Comparator): Patients will undergo bilateral RFA; the right side will be done following the traditional approach, and the left side will be done following the parasagittal approach. Traditional approach is done by placing the electrode at a 20 degrees' ipsilateral oblique angle to the sagittal plane toward the junction of the superior articular process and transverse process of the vertebral body to target the traversing medial branch nerve. The reason for the proposed angle is to avoid the mamillo-accessory ligament that may be ossified in up to 10% of the normal spine and potentially prevent proper coagulation of the medial branch nerve during the RFA procedure. Parasagittal (new) approach: is performed by placing the RF cannula parasagittally and more dorsally. To achieve maximum nerve coagulation, the electrode should be placed as parallel to the nerve as possible, and placing it parasagittally helps achieve this goal. The remainder of the procedure does not differ from the traditional method.
  Interventions: Procedure: Radiofrequency ablation of lumbar medial branch nerves.
- Subjects with traditional approach on the left side and parasagittal approach on the right side. (Active Comparator): Patients will undergo bilateral RFA; the left side will be done following the traditional approach, and the right side will be done following the parasagittal approach. Traditional approach is done by placing the electrode at a 20 degrees' ipsilateral oblique angle to the sagittal plane toward the junction of the superior articular process and transverse process of the vertebral body to target the traversing medial branch nerve. The reason for the proposed angle is to avoid the mamillo-accessory ligament that may be ossified in up to 10% of the normal spine and potentially prevent proper coagulation of the medial branch nerve during the RFA procedure. Parasagittal (new) approach: is performed by placing the RF cannula parasagittally and more dorsally. To achieve maximum nerve coagulation, the electrode should be placed as parallel to the nerve as possible, and placing it parasagittally helps achieve this goal. The remainder of the procedure does not differ from the traditional method.
  Interventions: Procedure: Radiofrequency ablation of lumbar medial branch nerves.

INTERVENTIONS:
Procedure: Radiofrequency ablation of lumbar medial branch nerves. — Traditional approach:
  The electrode is introduced at a 15-20 degrees' ipsilateral oblique angle to the sagittal plane toward the junction of the superior articular process (SAP) and transverse process (TP) of the vertebral body to target the traversing medial branch nerve.
  Parasagittal (new) approach:
  The RF cannula is placed parasagittally and more dorsally. The remainder of the procedure does not differ from the traditional method.

SUMMARY:
The purpose of this voluntary research study is to determine whether the parasagittal approach to lumbar medial branch (LMB) nerve radio frequency ablation (RFA) will have greater efficacy than the traditional approach to lumbar medial branch nerve radio frequency ablation.

DETAILED DESCRIPTION:
To determine whether the parasagittal approach to lumbar medial branch (LMB) nerve radiofrequency ablation (RFA) will have greater efficacy than the traditional approach to lumbar medial branch nerve radiofrequency ablation.

This will be accomplished by comparing the results between the newly proposed parasagittal approach and the traditional approach of medial branch RFA done on the same patient (different sites) with bilateral low back pain (LBP).

Traditional approach:

The electrode is introduced at a 15-20 degrees' ipsilateral oblique angle to the sagittal plane toward the junction of the superior articular process (SAP) and transverse process (TP) of the vertebral body to target the traversing medial branch nerve. The reason for the proposed angle is to avoid the mamillo-accessory ligament (MAL) that may be ossified in up to 10% of the normal spine and, in such cases, potentially prevent proper coagulation of the medial branch nerve during the RFA procedure.

Parasagittal (new) approach:

Recently, Tran et al. showed that MAL is located more dorsally than it was thought earlier and, therefore, can't interfere with nerve coagulation during the RFA. Consequently, they proposed abandoning the 20-degree angle used for the traditional approach and placing the radiofrequency cannula parasagittally and more dorsally. It is proposed that, in order to achieve maximum nerve coagulation, the electrode should be placed as parallel to the nerve as possible, and placing it parasagittally helps achieve this goal. The remainder of the procedure does not differ from the traditional method.

ELIGIBILITY:
Inclusion Criteria:

1. Bilateral equally intense axial low back pain
2. Pain duration of ≥ 6 months
3. Three-day average NRS scores of ≥ 3/10
4. Age greater than 18 years
5. Failure of conservative treatment, including nonsteroidal anti-inflammatory medications and physical therapy
6. Positive response to a series of two bilateral diagnostic lumbar medial branch nerve blocks (≥ 80% pain relief). This is the current standard of care.

Exclusion Criteria:

1. Radicular pain below the knee
2. Systemic infection or localized infection at the anticipated introducer entry site
3. Pregnancy
4. Allergy to Lidocaine
5. Bleeding dyscrasias
6. Patients unable to give informed consent
7. History of lumbar spine surgery at the affected levels
8. History of previous bilateral lumbar RFA of medial branches within the past six months.
9. Significant comorbid somatization or widespread pain with central sensitization
10. Secondary gain identified due to ongoing legal proceedings or worker's compensation
11. Cognitive impairment
12. Any pre-existing condition at the discretion of the provider that may confound interpretation of results -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
The number of patients whose procedure was successful (gained 50% or more reduction in numeric rating pain (NRS) scores). | Baseline
  The patients will describe the pain intensity using NRS - 11-point numeric rating scale, with 0 means no pain, and 10 - the worst possible pain intensity.
The number of patients whose procedure was successful (gained 50% or more reduction in numeric rating pain (NRS) scores). | 1 month post-procedure.
  The patients will describe the pain intensity using NRS - 11-point numeric rating scale, with 0 means no pain, and 10 - the worst possible pain intensity.
The number of patients whose procedure was successful (gained 50% or more reduction in numeric rating pain (NRS) scores). | 6 months post-procedure.
  The patients will describe the pain intensity using NRS - 11-point numeric rating scale, with 0 means no pain, and 10 - the worst possible pain intensity.

SECONDARY OUTCOMES:
Oswestry Disability index (ODI) | Baseline
  10 questions assessing the functional impairment by the pain, using a 50 point scale, with 0 meaning no disability, and 50 meaning complete disability.
Oswestry Disability index (ODI) | 1 month post-procedure.
  10 questions assessing the functional impairment by the pain, using a 50 point scale, with 0 meaning no disability, and 50 meaning complete disability.
Oswestry Disability index (ODI) | 6 months post-procedure.
  10 questions assessing the functional impairment by the pain, using a 50 point scale, with 0 meaning no disability, and 50 meaning complete disability.

OTHER OUTCOMES:
Number of subjects who ceased requiring analgesia | Baseline
  The patients will self-report their analgesic consumption.
Number of subjects who ceased requiring analgesia | 1 month post-procedure
  The patients will self-report their analgesic consumption.
Number of subjects who ceased requiring analgesia | 6 months post-procedure
  The patients will self-report their analgesic consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Yakov Vorobeychik, MD PhD, Principal Investigator — Professor, Department of Anesthesiology
Locations (1):
- Penn State Hershey College of Medicine, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD data that underlie the results reported in this article, after deidentification (text, tables, figures)
Supporting Information: Study Protocol
Time Frame: Beginning 1 month and ending 3 years following article publication.
Access Criteria: Researches who provide a methodologically sound proposal to achieve aims in the approved proposal. proposals should be directed to yvorobeychik@pennstatehealth.psu.edu.